CLINICAL TRIAL: NCT06089967
Title: Prospective Study to Evaluate Immune-Related Adverse Events and Associated Biomarkers in Patients Receiving Cancer Immunotherapy
Brief Title: Immune-Related Adverse Events and Associated Biomarkers in Patients Receiving Cancer Immunotherapy
Acronym: IMBARC
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00109576
Record Dates: First submitted 2023-10-11; First posted 2023-10-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Immune-related Adverse Event
Keywords: immunotherapy; immune-related adverse events; immune checkpoint inhibitors; immuno-oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Collection of blood, body fluids, and tissue for research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immune checkpoint inhibitor treatment: Adult cancer patients starting standard of care immune checkpoint inhibitor therapy. Participants willing to provide biospecimens (blood, body fluids and/or tissue) for research purposes. Participants will be followed for samples, irAEs and clinical data for up to one year after the end of treatment.
  Interventions: Other: Medical chart review

INTERVENTIONS:
Other: Medical chart review — Clinical data for all enrolled patients will be abstracted from the electronic medical record. This will include but will not be limited to patient demographics, primary disease (site, histology, histologic grade, staging system used, staging, molecular markers), prior cancer treatment, immunotherapy received, time of onset, treatment received for irAEs, and disease response to treatment. Clinical data will be collected for up to one year after discontinuation of cancer immunotherapy treatment.

SUMMARY:
The purpose of this project is to collect body samples like blood and tissue and health information from people receiving immune-based treatment for cancer. The body samples and health information will be stored for future research to understand more about side effects related to immune-based treatments for cancer.

DETAILED DESCRIPTION:
This is a prospective biospecimen and clinical data collection study in adult participants with melanoma, cutaneous squamous cell carcinoma, Merkel cell carcinoma, basal cell carcinoma, non-small cell lung cancer, small cell lung cancer, renal cell carcinoma, urothelial cancer, Hodgkins lymphoma, follicular lymphoma, head and neck carcinoma, hepatocellular carcinoma, breast carcinoma, gastric carcinoma, esophageal carcinoma, cholangiocarcinoma, pancreatic cancer, and any microsatellite instability-high (MSI-H) malignancy who are being treated with any of the following therapies alone or in combination:

* anti-PD-1 (nivolumab, pembrolizumab, cemiplimab)
* anti-CTLA-4 (ipilimumab or tremelimumab)
* anti-PD-L1 (atezolizumab, durvalumab, avelumab)
* anti-LAG3 (relatlimab)

Additional agents with similar mechanisms of action, e.g., targeting any of the above proteins may be included. Those with other targets may be considered on a case-by-case basis.

The goal of this study is to collect patient specimens from time points before, during, and after cancer immunotherapy discontinuation. Participants must agree to collection of biospecimens and clinical data. Biospecimens to be collected under this study include but are not limited to, blood specimens, primary or metastatic tumor specimen(s), end organ biospecimens such as bronchoalveolar/synovial fluid or colon tissues biopsies, and any other tissues that are biopsied for evaluation of a potential immune-related adverse events (irAE). Clinical data, including, but not limited to, cancer diagnosis, staging, treatment, toxicities and management, will be collected for up to one year after discontinuation of cancer immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Selected for standard of care therapy with a checkpoint inhibitor or immunotherapeutic as recommended by their medical oncologist, including but not limited to: pembrolizumab, nivolumab, cemiplimab, ipilimumab, tremelimumab, durvalumab, atezolizumab, avelumab, and relatlimab.
3. Histologically confirmed diagnosis with a malignancy, including but not limited to: melanoma, cutaneous squamous cell carcinoma, Merkel cell carcinoma, basal cell carcinoma, non-small cell lung cancer, small cell lung cancer, renal cell carcinoma, urothelial cancer, Hodgkins lymphoma, follicular lymphoma, head and neck carcinoma, hepatocellular carcinoma, breast carcinoma, gastric carcinoma, esophageal carcinoma, cholangiocarcinoma, pancreatic cancer, and any microsatellite instability-high (MSI-H) malignancy.
4. Legally be allowed to sign as well as be able to understand and date the study and written informed consent to take part in all mentioned evaluations.

Exclusion Criteria:

1. Cytotoxic chemotherapy or biologic agents (eg. cytokines or antibodies) within 4 weeks of treatment initiation.
2. Steroids equivalent to or greater than prednisone 10 mg daily within 2 weeks of treatment initiation.
3. Antibiotic therapies within 2 weeks of treatment initiation.
4. Previously confirmed diagnosis of an autoimmune disease felt by the investigators to complicate data analysis. Those autoimmune conditions generally felt to be benign such as atopic dermatitis will be considered for enrollment on a case-by-case basis.
5. Organ transplant recipients on immunosuppressive agents.
6. Immunosuppressive drugs in the last 12 weeks for reasons other than autoimmune disease or organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients at Duke University Health Systems starting immune checkpoint inhibitor therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Number of participants cancer patients with immune-related adverse events with biospecimens and clinical data collected | Up to 1 year after the end of immune checkpoint inhibitor therapy
  Clinical database of participants receiving immune checkpoint inhibitors paired with biospecimen collection.
  Participant specimens are collected at time points before, during, and after cancer immunotherapy discontinuation. Clinical data collection includes, but is not limited to patient demographics, primary disease (site, histology, histologic grade, staging system used, staging, molecular markers), prior cancer treatment, immunotherapy received, time of onset, treatment received for irAEs, and disease response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Hanks, MD PhD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No